CLINICAL TRIAL: NCT01547299
Title: A Randomized, Open-label, Phase 2 Study Of Mdv3100 As A Neoadjuvant Therapy For Patients Undergoing Prostatectomy For Localized Prostate Cancer
Brief Title: Study of Enzalutamide (Formerly MDV3100) as a Neoadjuvant Therapy for Patients Undergoing Prostatectomy for Localized Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Astellas Pharma Inc (Industry); Medivation LLC, a wholly owned subsidiary of Pfizer Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDV3100-07; C3431019 (Other: Alias Study Number)
Record Dates: First submitted 2012-02-27; First posted 2012-03-07 (Estimated); Results first posted 2015-04-10 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; prostatectomy; neoadjuvant
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; Leuprolide; Dutasteride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enzalutamide alone (Experimental): Enzalutamide 160 mg, orally, once daily
  Interventions: Drug: Enzalutamide
- Enzalutamide & Leuprolide & Dutasteride (Experimental): Enzalutamide 160 mg, orally, once daily and leuprolide 22.5 mg, intramuscular injection, every 3 months, and dutasteride, 0.5 mg, orally, once daily
  Interventions: Drug: Enzalutamide; Drug: Leuprolide; Drug: Dutasteride

INTERVENTIONS:
Drug: Enzalutamide
  Other Names: MDV3100
Drug: Leuprolide
  Arms: Enzalutamide & Leuprolide & Dutasteride
Drug: Dutasteride
  Arms: Enzalutamide & Leuprolide & Dutasteride

SUMMARY:
The purpose of this study is to determine if enzalutamide is an effective therapy in treating localized prostate cancer prior to prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide informed consent
* 18 years of age or older
* Histologically confirmed adenocarcinoma of the prostate
* Must be a candidate for radical prostatectomy and considered surgically resectable

Exclusion Criteria:

* Stage T4 prostate cancer by clinical or radiologic evaluation
* Treatment with an investigational agent within 4 weeks prior to randomization
* Received therapy for other neoplastic disorders within 5 years
* Hypogonadism or severe androgen deficiency

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 52 (Actual)
Dates: Start 2012-03-31 (Actual); Primary Completion 2013-11-30 (Actual); Study Completion 2013-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (2):
  - Boston, Massachusetts
  - Seattle, Washington
- Canada (2):
  - Vancouver, British Columbia
  - Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

RESULTS

PARTICIPANT FLOW:
Groups:
- Enzalutamide + Leuprolide + Dutasteride: Participants were administered 160 milligram (mg) of Enzalutamide orally once daily, 22.5 mg of Leuprolide every 3 months through intramuscular injection and 0.5 mg of Dutasteride orally once daily for up to 180 days.
- Enzalutamide: Participants were administered 160 mg of Enzalutamide orally once daily for up to 180 days.
Period: Overall Study
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Started | 25 | 27
Completed | 23 | 25
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Enzalutamide + Leuprolide + Dutasteride: Participants were administered 160 mg of Enzalutamide orally once daily, 22.5 mg of Leuprolide every 3 months through intramuscular injection and 0.5 mg of Dutasteride orally once daily for up to 180 days.
- Total: Total of all reporting groups
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (6.95) | 61.4 (7.65) | 61.1 (7.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 25 | 27 | 52

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Complete Response Rate
Description: Pathologic complete response rate was defined as percentage of participants with pathologic complete response. Pathologic complete response rate following triplet therapy (enzalutamide in combination with leuprolide and dutasteride) and enzalutamide alone when administered as neoadjuvant therapy for 180 days prior to prostatectomy in participants with localized prostate cancer. Pathologic complete response was defined as the absence of morphologically identifiable carcinoma in the prostatectomy specimen, as assessed by the local and central pathologist.
Time Frame: Day 180
Population: All participants randomly assigned to study treatment (intent-to-treat population) with a prostatectomy sample evaluated by the local and central pathologist. Here, "N" signifies number of participants evaluable for this specified outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Number analyzed (Participants) | 23 | 25
percentage of participants
  Local pathologist | 8.7 [1.1 to 28.0] | 0.0 [0.0 to 13.7]
  Central pathologist | 4.3 [0.1 to 21.9] | 0.0 [0.0 to 13.7]

2. Secondary Outcome: Percentage of Participants With Positive Surgical Margins
Description: To determine the percentage of participants with positive surgical margins at prostatectomy as assessed by the local and central pathologist. Surgical margin, also known as tumor free margin referred to the visible normal tissue or skin margin that was removed with the surgical excision of a tumor, growth, or malignancy. The margin was described as positive when the pathologist finds cancer cells at the edge of the tissue, suggesting that all of the cancer has not been removed.
Time Frame: Day 180
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Number analyzed (Participants) | 23 | 25
percentage of participants
  Local pathologist | 4.3 [0.1 to 21.9] | 12.0 [2.5 to 31.2]
  Central pathologist | 21.7 [7.5 to 43.7] | 16.0 [4.5 to 36.1]

3. Secondary Outcome: Percentage of Participants With Extracapsular Extension: Local Review
Description: To determine the percentage of participants with extracapsular extension at prostatectomy as assessed by the local pathologist. Extracapsular extension was defined as prostate cancer cells when extended into the prostate capsule or outer lining of the prostate gland.
Time Frame: Day 180
Population: All participants randomly assigned to study treatment (intent-to-treat population) with a prostatectomy sample evaluated by the local pathologist. Here, "N" signifies number of participants evaluable for this specified outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Number analyzed (Participants) | 23 | 25
percentage of participants | 26.1 [10.2 to 48.4] | 36.0 [18.0 to 57.5]

4. Secondary Outcome: Percentage of Participants With Extracapsular Extension: Central Review
Description: To determine the percentage of participants with extracapsular extension at prostatectomy as assessed by the central pathologist. Extracapsular extension was defined as prostate cancer cells when extended into the prostate capsule or outer lining of the prostate gland.
Time Frame: Day 180
Population: All participants randomly assigned to study treatment with a prostatectomy sample evaluated by the central pathologist. One participant in the Enzalutamide treatment arm was excluded from the analysis because the result reported by the central lab was indeterminate. Here, "N" signifies number of participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Number analyzed (Participants) | 23 | 24
percentage of participants | 56.5 [34.5 to 76.8] | 70.8 [48.9 to 87.4]

5. Secondary Outcome: Percentage of Participants With Positive Seminal Vesicles
Description: To determine the percentage of participants with positive seminal vesicles at prostatectomy as assessed by the local and central pathologist. Seminal vesicles or seminal glands, were defined as a pair of simple tubular glands located within the pelvis. They secrete fluid that partly composes the semen. Seminal vesicles with cancer cells in them were called positive seminal vesicles.
Time Frame: Day 180
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Number analyzed (Participants) | 23 | 25
percentage of participants
  Local pathologist | 30.4 [13.2 to 52.9] | 36.0 [18.0 to 57.5]
  Central pathologist | 30.4 [13.2 to 52.9] | 36.0 [18.0 to 57.5]

6. Secondary Outcome: Percentage of Participants With Positive Lymph Nodes
Description: To determine the percentage of participants with positive lymph nodes at prostatectomy as assessed by the local and central pathologist. Lymph nodes were small clumps of immune cells that act as filters for the lymphatic system. Lymph nodes with cancer cells in them were called positive lymph nodes.
Time Frame: Day 180
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Number analyzed (Participants) | 23 | 25
percentage of participants
  Local pathologist | 26.1 [10.2 to 48.4] | 4.0 [0.1 to 20.4]
  Central pathologist | 26.1 [10.2 to 48.4] | 4.0 [0.1 to 20.4]

7. Secondary Outcome: Prostate-Specific Antigen (PSA) Nadir
Description: To determine the effects on PSA as measured by the lowest post baseline PSA value prior to prostatectomy. Prostate-specific antigen (PSA) was a protein produced by normal, as well as malignant, cells of the prostate gland. The PSA nadir was the participant's lowest observed post baseline PSA value.
Time Frame: Day 195
Population: All participants randomly assigned to study treatment (intent-to-treat population) with a baseline PSA and at least one post baseline PSA. Here, "N" signifies number of participants evaluable for this specified outcome measure.
Measure: Median (Full Range); unit: microgram per liter (mcg/L)
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Number analyzed (Participants) | 24 | 25
microgram per liter (mcg/L) | 0.04 [0.01 to 0.53] | 0.51 [0.02 to 8.80]

8. Secondary Outcome: Time to Prostate-Specific Antigen (PSA) Nadir
Description: To determine the effects on PSA as measured by the time to the lowest post baseline PSA value prior to prostatectomy. Prostate-specific antigen (PSA) was a protein produced by normal, as well as malignant, cells of the prostate gland. The PSA nadir was the participant's lowest observed post baseline PSA value.
Time Frame: Day 195
Population: All participants randomly assigned to study treatment (intent-to-treat population) with a baseline PSA and at least one post baseline PSA.
Measure: Median (Full Range); unit: days
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Number analyzed (Participants) | 25 | 27
days | 5.09 [2.79 to 6.44] | 6.01 [2.89 to 6.64]

9. Secondary Outcome: Percentage of Participants With Reduction in Prostate-Specific Antigen (PSA)
Description: To determine the effects on PSA as measured by the percentage of participants with PSA less than (<) 0.2 nanogram per milliliter (ng/mL), and a 50 percent (%) and 90% decrease in PSA value prior to prostatectomy. Prostate-specific antigen (PSA) was a protein produced by normal, as well as malignant, cells of the prostate gland.
Time Frame: Day 195
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Number analyzed (Participants) | 25 | 27
percentage of participants
  PSA < 0.2 ng/mL | 92.0 [74.0 to 99.0] | 29.6 [13.8 to 50.2]
  50% decrease in PSA | 100.0 [86.3 to 100.0] | 100.0 [87.2 to 100.0]
  90% decrease in PSA | 100.0 [86.3 to 100.0] | 63.0 [42.4 to 80.6]

10. Secondary Outcome: Health-Related Quality of Life (HRQoL): Number of Participants With The Expanded Prostate Cancer Index Composite (EPIC) Sexual Domain Summary Score
Description: EPIC sexual domain was HRQoL instrument that measured the effects of prostate cancer treatment on a participant's sexual function and sexual satisfaction. Sexual domain summary score was measured on a scale ranged from 0 (worst) to 100 (best) with higher scores representing better sexual function and satisfaction. Best change from baseline category in EPIC sexual domain summary score ranged from worsened to improved where worsened indicated decrease of at least 1 minimally important difference, stable indicated changed by less than 1 minimally important difference and improved indicated increase of at least 1 minimally important difference. Minimally important difference was defined as one-half of the standard deviation of baseline score. Number of participants within each category are reported below.
Time Frame: Day 180
Population: All participants randomly assigned to study treatment (intent-to-treat population) with a baseline and at least one post baseline score. Here, "N" signifies number of participants evaluable for this specified outcome measure.
Measure: Number; unit: participants
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Number analyzed (Participants) | 16 | 16
participants
  Worsened | 11 | 10
  Stable | 4 | 6
  Improved | 1 | 0

11. Secondary Outcome: Health-Related Quality of Life (HRQoL): Number of Participants With Expanded Prostate Cancer Index Composite (EPIC) Sexual Function Subscale Score
Description: EPIC sexual function subscale was HRQoL instrument that measured the effects of prostate cancer treatment on a participant's sexual function and sexual satisfaction. EPIC sexual function subscale was a component of sexual domain that was evaluated on a distinct set of questions. It was measured on a scale ranged from 0 (worst) to 100 (best) with higher scores representing better sexual function. Best change from baseline category in EPIC sexual function subscale score ranged from worsened to improved where worsened indicated decrease of at least 1 minimally important difference, stable indicated changed by less than 1 minimally important difference and improved indicated increase of at least 1 minimally important difference. Minimally important difference was defined as one-half of the standard deviation of baseline score. Number of participants within each category are reported below.
Time Frame: Day 180
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Number analyzed (Participants) | 15 | 17
participants
  Worsened | 11 | 12
  Stable | 4 | 5
  Improved | 0 | 0

12. Secondary Outcome: Health-Related Quality of Life (HRQoL): Number of Participants With Expanded Prostate Cancer Index Composite (EPIC) Sexual Bother Subscale Score
Description: EPIC sexual bother subscale was HRQoL instrument that measured the effects of prostate cancer treatment on a participant's sexual function and sexual satisfaction. EPIC sexual bother subscale was a component of sexual domain that was evaluated on a distinct set of questions. It was measured on a scale ranged from 0 (worst) to 100 (best) with higher scores representing less sexual bother and difficulty. Best change from baseline category in EPIC sexual bother subscale score ranged from worsened to improved where worsened indicated decrease of at least 1 minimally important difference, stable indicated changed by less than 1 minimally important difference and improved indicated increase of at least 1 minimally important difference. Minimally important difference was defined as one-half of the standard deviation of baseline score. Number of participants within each category are reported below.
Time Frame: Day 180
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Number analyzed (Participants) | 16 | 16
participants
  Worsened | 7 | 5
  Stable | 9 | 7
  Improved | 0 | 4

13. Secondary Outcome: Health-Related Quality of Life (HRQoL): Number of Participants With Expanded Prostate Cancer Index Composite (EPIC) Hormonal Domain Summary Score
Description: EPIC Hormonal Domain was HRQoL instrument that measured the effects of prostate cancer treatment on a participant's hormonal function. It was measured on a scale ranged from 0 (worst) to 100 (best) scale with higher scores representing better hormonal function. Best change from baseline category in EPIC hormonal domain summary score ranged from worsened to improved where worsened indicated decrease of at least 1 minimally important difference, stable indicated changed by less than 1 minimally important difference and improved indicated increase of at least 1 minimally important difference. Minimally important difference was defined as one-half of the standard deviation baseline score. Number of participants within each category are reported below.
Time Frame: Day 180
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Number analyzed (Participants) | 16 | 18
participants
  Worsened | 10 | 10
  Stable | 3 | 7
  Improved | 3 | 1

14. Secondary Outcome: Health-Related Quality of Life (HRQoL): Number of Participants With Expanded Prostate Cancer Index Composite (EPIC) Hormonal Function Subscale Score
Description: EPIC hormonal function subscale score was HRQoL instrument that measured the effects of prostate cancer treatment on a participant's hormonal function. EPIC hormonal function subscale was a component of hormonal domain that was evaluated on a distinct set of questions. It was measured on a scale ranged from 0 (worst) to 100 (best) scale with higher scores representing better hormonal function. Best change from baseline category in EPIC hormonal function subscale score ranged from worsened to improved where worsened indicated decrease of at least 1 minimally important difference, stable indicated changed by less than 1 minimally important difference and improved indicated increase of at least 1 minimally important difference. Minimally important difference was defined as one-half of the standard deviation baseline score. Number of participants within each category are reported below.
Time Frame: Day 180
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Number analyzed (Participants) | 16 | 18
participants
  Worsened | 11 | 11
  Stable | 2 | 7
  Improved | 3 | 0

15. Secondary Outcome: Health-Related Quality of Life (HRQoL): Number of Participants With Expanded Prostate Cancer Index Composite (EPIC) Hormonal Bother Subscale Score
Description: EPIC hormonal bother subscale score was HRQoL instrument that measured the effects of prostate cancer treatment on a participant's hormonal function. EPIC hormonal bother subscale was a component of hormonal domain that was evaluated on a distinct set of questions. It was measured on a scale ranged from 0 (worst) to 100 (best) scale with higher scores representing less hormonal bothering. Best change from baseline category in EPIC hormonal bother subscale score ranged from worsened to improved where worsened indicated decrease of at least 1 minimally important difference, stable indicated changed by less than 1 minimally important difference and improved indicated increase of at least 1 minimally important difference. Minimally important difference was defined as one-half of the standard deviation baseline score. Number of participants within each category are reported below.
Time Frame: Day 180
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Number analyzed (Participants) | 16 | 18
participants
  Worsened | 9 | 6
  Stable | 5 | 11
  Improved | 2 | 1

16. Secondary Outcome: Health-Related Quality of Life (HRQoL): Number of Participants With Twelve-Item Short Form Version 2 General Health Domain Score
Description: The Twelve-Item Short Form Version 2 was HRQoL instrument that measured general health and well-being across physical and mental components. The general health domain score contained 1 item scored on a scale of 1 to 5 where 1=excellent to 5=poor health, where higher score indicated worse health status. Best change from baseline category in general health domain score ranged from worsened (decrease of at least 1 minimally important difference), stable (changed by less than 1 minimally important difference), or improved (increase of at least 1 minimally important difference). Minimally important difference was defined as one-half the standard deviation of the score of interest at baseline.
Time Frame: Day 180
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Number analyzed (Participants) | 16 | 18
participants
  Worsened | 5 | 5
  Stable | 9 | 6
  Improved | 2 | 7

17. Secondary Outcome: Health-Related Quality of Life (HRQoL): Number of Participants With Twelve-Item Short Form Version 2 Physical Functioning Domain Score
Description: The Twelve-Item Short Form Version 2 was HRQoL instrument that measured general health and well-being across physical and mental components. The physical functioning domain score contained 2 items each scored on a scale of 1 to 5 where 1=excellent physical functioning to 5=poor physical functioning. Physical functioning domain total score ranged from 1 to 10, where higher scores indicated poor physical functioning. Best change from baseline category in physical functioning domain score ranged from worsened (decrease of at least 1 minimally important difference), stable (changed by less than 1 minimally important difference), or improved (increase of at least 1 minimally important difference). Minimally important difference was defined as one-half the standard deviation of the score of interest at baseline.
Time Frame: Day 180
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Number analyzed (Participants) | 16 | 18
participants
  Worsened | 3 | 2
  Stable | 12 | 15
  Improved | 1 | 1

18. Secondary Outcome: Health-Related Quality of Life (HRQoL): Number of Participants With Twelve-Item Short Form Version 2 Role-Emotional Domain Score
Description: The Twelve-Item Short Form Version 2 was HRQoL instrument that measured general health and well-being across physical and mental components. The mental health domain score had 2 items scored on a scale of 1 to 5, where higher scores indicated worse mental status. The total score ranged from 1 to 10, where higher scores indicated worse mental status. Best change from baseline category in mental component summary ranged from worsened (decrease of at least 1 minimally important difference), stable (changed by less than 1 minimally important difference), or improved (increase of at least 1 minimally important difference). Minimally important difference was defined as one-half the standard deviation of the score of interest at baseline.
Time Frame: Day 180
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Number analyzed (Participants) | 16 | 18
participants
  Worsened | 3 | 1
  Stable | 9 | 10
  Improved | 4 | 7

19. Secondary Outcome: Health-Related Quality of Life (HRQoL): Number of Participants With Twelve-Item Short Form Version 2 Mental Component Summary
Description: The Twelve-Item Short Form Version 2 was HRQoL instrument that measured general health and well-being across physical and mental components. The mental health domain score had 2 items scored on a scale of 1 to 5 where for 1 item 1=all of the time person felt calm and peaceful to 5=none of the time person felt calm and peaceful. The score ranged from 1 to 5, where higher scores meant worse mental status. For other item 1=all of the time person felt downhearted and blue to 5=none of the time person felt downhearted and blue. The score ranged from 1 to 5, where higher scores meant better mental status. Best change from baseline category in mental component summary ranged from worsened (decrease of at least 1 minimally important difference), stable (changed by less than 1 minimally important difference), or improved (increase of at least 1 minimally important difference). Minimally important difference was defined as one-half the standard deviation of the score of interest at baseline.
Time Frame: Day 180
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Number analyzed (Participants) | 16 | 17
participants
  Worsened | 4 | 1
  Stable | 8 | 11
  Improved | 4 | 5

20. Secondary Outcome: Pharmacodynamic Effects: Tissue Dihydrotestosterone (DHT)
Description: To determine pharmacodynamic effects as measured by the amount of tissue DHT in prostatectomy specimens following radical prostatectomy.
Time Frame: Day 180
Population: All participants randomly assigned to study treatment (intent-to-treat population) with a prostatectomy sample evaluated by the central pathologist. Here, "N" signifies number of participants evaluable for this specified outcome measure.
Measure: Mean (Standard Deviation); unit: picogram per milligram
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Number analyzed (Participants) | 23 | 25
picogram per milligram | 0.04 (0.01) [0.02 to 0.06] | 3.34 (1.57) [0.86 to 8.92]

21. Secondary Outcome: Pharmacodynamic Effects: Tissue Testosterone
Description: To determine pharmacodynamic effects as measured by the amount of tissue testosterone in prostatectomy specimens following radical prostatectomy.
Time Frame: Day 180
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: picogram per milligram
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Number analyzed (Participants) | 23 | 25
picogram per milligram | 0.18 (0.13) [0.04 to 0.54] | 0.90 (0.86) [0.16 to 4.36]

22. Secondary Outcome: Pharmacodynamic Effects: Assessment of Apoptosis
Description: To determine the effects of triplet therapy and enzalutamide alone on apoptosis in prostatectomy specimens. Apoptosis was a process of biochemical events that lead to characteristic cell changes and death.
Time Frame: Day 180
Population: Data for this outcome measure was not collected as assessment of apoptosis was not performed due to limited amounts of tissue samples available.
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: Pharmacodynamic Effects: Assessment of Mitotic Index
Description: Assessment was performed to determine the effects of triplet therapy and enzalutamide alone on mitotic index. Mitotic index was defined as the ratio between the numbers of cells in a population undergoing mitosis to the number of cells in a population not undergoing mitosis in prostatectomy specimens.
Time Frame: Day 180
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Number analyzed (Participants) | 22 | 25
ratio | 0.9 (1.51) | 2.6 (2.81)

24. Secondary Outcome: Pharmacodynamic Effects: Assessment of Androgen Receptor Signaling as Measured by Intensity of Androgen Receptor Immunohistochemical (IHC) Staining
Description: To determine the effects of triplet therapy and enzalutamide alone on androgen receptor signaling in prostatectomy specimens. Androgen receptor (AR) was a type of nuclear receptor that was activated by binding either of the androgenic hormones, testosterone, or dihydrotestosterone in the cytoplasm and then translocating into the nucleus. Androgen receptor (AR) signaling represented the major therapeutic target for treating metastatic prostate cancer. Assessment of androgen receptor signaling was measured by intensity of androgen receptor IHC staining and were graded as 0 (absent), 1 (weak), 2 (moderate) and 3 (strong). Percentage of participants within each grade are reported below.
Time Frame: Day 180
Population: All participants randomly assigned to study treatment (intent-to-treat population) with a prostatectomy sample evaluated by the local pathologist.
Measure: Number; unit: percentage of participants
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Number analyzed (Participants) | 25 | 27
percentage of participants
  0 | 0.0 | 0.0
  1 | 5.6 | 0.0
  2 | 27.8 | 5.3
  3 | 66.7 | 94.7

25. Secondary Outcome: Serum Dihydrotestosterone (DHT): Baseline
Time Frame: Baseline
Population: All participants randomly assigned to study treatment (intent-to-treat population) with a baseline serum DHT result. Here, "N" signifies number of participants evaluable for this specified outcome measure.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Number analyzed (Participants) | 23 | 27
ng/mL | 0.34 [0.08 to 0.58] | 0.29 [0.16 to 0.85]

26. Secondary Outcome: Serum Dihydrotestosterone (DHT): Day 180
Time Frame: Day 180
Population: All participants randomly assigned to study treatment (intent-to-treat population) with 180 days post baseline serum DHT result. Here, "N" signifies number of participants evaluable for this specified outcome measure.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Number analyzed (Participants) | 25 | 25
ng/mL | 0.01 [0.01 to 0.04] | 0.51 [0.10 to 1.10]

27. Secondary Outcome: Change From Baseline in Serum Dihydrotestosterone (DHT) at Day 180
Description: To determine serum hormone effects as measured by change in DHT values from baseline to the completion of therapy.
Time Frame: Day 180
Population: All participants randomly assigned to study treatment (intent-to-treat population) with a serum DHT result at baseline and 180 days post baseline. Here, "N" signifies number of participants evaluable for this specified outcome measure.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Number analyzed (Participants) | 23 | 25
ng/mL | -0.33 [-0.57 to -0.07] | 0.25 [-0.16 to 0.71]

28. Secondary Outcome: Serum Testosterone: Baseline
Time Frame: Baseline
Population: All participants randomly assigned to study treatment (intent-to-treat population) with a baseline serum testosterone result. Here, "N" signifies number of participants evaluable for this specified outcome measure.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Number analyzed (Participants) | 23 | 27
ng/mL | 4.10 [0.77 to 6.77] | 3.69 [2.00 to 7.91]

29. Secondary Outcome: Serum Testosterone: Day 180
Time Frame: Day 180
Population: All participants randomly assigned to study treatment (intent-to-treat population) with a 180 days post baseline serum testosterone result. Here, "N" signifies number of participants evaluable for this specified outcome measure.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Number analyzed (Participants) | 25 | 25
ng/mL | 0.12 [0.05 to 0.29] | 9.76 [1.99 to 16.63]

30. Secondary Outcome: Change From Baseline in Serum Testosterone at Day 180
Description: To determine serum hormone effects as measured by change in testosterone at baseline and at completion of therapy.
Time Frame: Day 180
Population: All participants randomly assigned to study treatment (intent-to-treat population) with a serum testosterone result at baseline and 180 days post baseline. Here, "N" signifies number of participants evaluable for this specified outcome measure.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Number analyzed (Participants) | 23 | 25
ng/mL | -4.00 [-6.67 to -0.67] | 5.74 [-1.94 to 12.29]

31. Secondary Outcome: Number of Participants With Adverse Events (AEs) That Led to Dose Interruption, Dose Reduction, and Study Drug Discontinuation
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: From baseline up to 210 days
Population: All participants who received at least 1 partial dose of enzalutamide (safety population).
Measure: Number; unit: participants
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Number analyzed (Participants) | 25 | 27
participants
  Permanent Discontinuation of Enzalutamide | 0 | 0
  Temporary Interruption of Enzalutamide | 3 | 0
  Dose Reduction of Enzalutamide | 0 | 0
  Study Drug Discontinuation | 0 | 0

ADVERSE EVENTS:
Time Frame: From baseline to 30 days after the last dose of study drug, up to 210 days.
Description: Same event may appear as AE and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another or 1 participant may have experienced both serious and non-serious event during study. Safety data set included all participants who received at least one partial dose of study drug.
Arm/Group | Enzalutamide + Leuprolide + Dutasteride | Enzalutamide
Serious Adverse Events (participants affected / at risk) | 3/25 | 2/27
Other Adverse Events (participants affected / at risk) | 25/25 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enzalutamide + Leuprolide + Dutasteride (N=25) | Enzalutamide (N=27)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
Pelvic abscess (Infections and infestations) | 0 | 1
Clostridial infection (Infections and infestations) | 1 | 0
Lymphocele (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Enzalutamide + Leuprolide + Dutasteride (N=25) | Enzalutamide (N=27)
Fatigue (General disorders) | 15 | 19
Hot flush (Vascular disorders) | 24 | 7
Gynaecomastia (Reproductive system and breast disorders) | 3 | 17
Insomnia (Psychiatric disorders) | 9 | 6
Libido decreased (Psychiatric disorders) | 8 | 4
Breast tenderness (Reproductive system and breast disorders) | 2 | 9
Diarrhoea (Gastrointestinal disorders) | 6 | 5
Pollakiuria (Renal and urinary disorders) | 6 | 4
Incision site pain (Injury, poisoning and procedural complications) | 4 | 5
Erectile dysfunction (Reproductive system and breast disorders) | 2 | 6
Breast pain (Reproductive system and breast disorders) | 0 | 7
Urinary incontinence (Renal and urinary disorders) | 2 | 5
Constipation (Gastrointestinal disorders) | 4 | 2
Headache (Nervous system disorders) | 3 | 3
Hypertension (Vascular disorders) | 3 | 3
Incontinence (Renal and urinary disorders) | 3 | 3
Memory impairment (Nervous system disorders) | 3 | 3
Nasopharyngitis (Infections and infestations) | 4 | 2
Nausea (Gastrointestinal disorders) | 4 | 2
Restless leg syndrome (Nervous system disorders) | 3 | 3
Anxiety (Psychiatric disorders) | 4 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Nipple pain (Reproductive system and breast disorders) | 1 | 3
Nocturia (Renal and urinary disorders) | 3 | 1
Oedema peripheral (General disorders) | 2 | 2
Pyrexia (General disorders) | 2 | 2
Sinusitis (Infections and infestations) | 3 | 1
Urinary tract infection (Infections and infestations) | 3 | 1
Amnesia (Nervous system disorders) | 0 | 3
Chills (General disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Depression (Psychiatric disorders) | 2 | 1
Diverticulitis (Infections and infestations) | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2
Mental impairment (Nervous system disorders) | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Oestradiol increased (Investigations) | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Weight decreased (Investigations) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood creatinine increased (Investigations) | 0 | 2
Dysuria (Renal and urinary disorders) | 0 | 2
Haematochezia (Gastrointestinal disorders) | 0 | 2
Micturition urgency (Renal and urinary disorders) | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Penile pain (Reproductive system and breast disorders) | 2 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2
Urinary retention (Renal and urinary disorders) | 0 | 2
Weight increased (Investigations) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI agrees not to independently publish the results before the publication of the multi-center PI paper. Sponsor shall review and comment 30 days prior to submission or disclosure. If publication or disclosure contains Sponsor Confidential Information, other than study data, PI agrees to remove Confidential Information from publication or disclosure. Sponsor may request that PI delay such publication for an additional 60 days to protect the patentability of any invention described.